CLINICAL TRIAL: NCT02797665
Title: Treatment of Obstructive Jaundice in Autoimmune Pancreatitis and/or Immunoglobulin G4-related Sclerosing Cholangitis by Corticosteroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-844
Record Dates: First submitted 2016-06-06; First posted 2016-06-13 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Autoimmune Pancreatitis; IgG4-related Sclerosing Cholangitis; Obstructive Jaundice
MeSH Terms: conditions — Autoimmune Pancreatitis; Jaundice, Obstructive | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Steroids group (Active Comparator): The patients will be treated with oral corticosteroids (prednisone 0.6mg/kg/d) alone.
  Interventions: Drug: corticosteroids
- Stent group (Active Comparator): The patients will be treated with oral corticosteroids and biliary stent.
  Interventions: Drug: corticosteroids; Procedure: biliary stent

INTERVENTIONS:
Drug: corticosteroids — prednisone 0.6mg/kg/d
Procedure: biliary stent — placement of biliary stent during endoscopic retrograde cholangiopancreatography (ERCP)
  Arms: Stent group

SUMMARY:
This study evaluates corticosteroids in the treatment of obstructive jaundice in autoimmune pancreatitis and/or immunoglobulin G4 (IgG4)-related sclerosing cholangitis in adults. Half of participants will receive corticosteroids alone, while the other half will receive corticosteroids with biliary stent at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* adults greater than 18 years-old;
* autoimmune pancreatitis and/or IgG4-related sclerosing cholangitis;
* obstructive jaundice

Exclusion Criteria:

* malignancies; active infections;
* pregnancy or breast feeding;
* standard contraindications to ERCP;
* unwillingness or inability to consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate of obstructive jaundice | Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Yang, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China